CLINICAL TRIAL: NCT00000408
Title: Evaluation of a Low Back Pain Patient Education Program
Brief Title: Low Back Pain Patient Education Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kate Lorig, professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR044939 (NIH); R01AR044939 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2003-02

CONDITIONS: Low Back Pain
Keywords: Health education; Back injury; Chronic pain; Education/evaluation planning; Outcomes research
MeSH Terms: conditions — Low Back Pain; Health Education; Back Injuries; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- email discussion group (Experimental)
  Interventions: Procedure: Patient education evaluation
- rancomized control group (No Intervention): usual care

INTERVENTIONS:
Procedure: Patient education evaluation
  Arms: email discussion group

SUMMARY:
Back pain is one of the most common of all symptoms. It is also a great cause of days lost from work and visits to health care providers. This study will develop and evaluate an approach to low back pain that allows subjects to talk with each other and with health professionals via an Internet discussion group. Results we will look at include health behaviors, such as exercise; health status, such as pain and disability; and health care use, such as number of visits to doctors and other health care providers. Anyone 18 years old or older who lives in the United States and has ongoing Internet access can take part in the study. All subjects must have back pain and meet the eligibility criteria listed below.

DETAILED DESCRIPTION:
This study will develop and evaluate in a randomized trial a low back pain intervention that allows subjects to talk with each other and with health professionals via an Internet discussion group. The intervention consists of a book and a videotape and is based on interaction with other participants in the program and health professionals through a closed password protected moderated Internet discussion group. Outcome measures include health behaviors, such as exercise; health status, such as pain and disability; and health care use, such as number of visits to doctors and other health care providers. Patients will be randomized either to the treatment group and followed for 6, 12, 18, and 24 months with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must live in the United States
* Must understand and write English
* Must have access to a computer with e-mail and expect to have this access for at least 3 years
* Must be 18 years old
* Must have seen a doctor for back pain at least once in the past year

Exclusion Criteria:

* Pregnancy
* Back surgery in the past 6 months
* Expectation of having back surgery in the next 6 months
* Back pain due to a car accident or other major injury within the last 6 months
* Back pain or sciatica due to systemic disease (inflammatory rheumatic diseases, tumor, or other)
* Major physical or mental health condition for which one is currently being treated that severely limits daily activities
* Terminal illness
* Receiving disability or workers compensation insurance payments for back pain or sciatica
* Presently involved in legal proceedings because of back pain or sciatica
* Difficulty with bladder or bowel control that began with back pain or sciatica
* No visits to a doctor in the past year for back pain or sciatica
* Numbness in crotch area that began with back pain or sciatica
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 1998-02; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate R. Lorig, Dr.P.H., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Result] Lorig KR, Laurent DD, Deyo RA, Marnell ME, Minor MA, Ritter PL. Can a Back Pain E-mail Discussion Group improve health status and lower health care costs?: A randomized study. Arch Intern Med. 2002 Apr 8;162(7):792-6. doi: 10.1001/archinte.162.7.792. PMID 11926853
- [Result] Bruce B, Lorig K, Laurent D, Ritter P. The impact of a moderated e-mail discussion group on use of complementary and alternative therapies in subjects with recurrent back pain. Patient Educ Couns. 2005 Sep;58(3):305-11. doi: 10.1016/j.pec.2004.08.012. PMID 16122642